CLINICAL TRIAL: NCT07002671
Title: The Significance of Preoperatively Calculated HALP Score in Differentiating Complicated Acute Appendicitis in Patients With Acute Appendicitis
Brief Title: The Role of Preoperative HALP Score in Differentiating Complicated Acute Appendicitis
Acronym: Appendicitis
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Associate, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: 2025/9-8
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Appendicitis; Acute Appendicitis Without Peritonitis; Acute Appendicitis With Appendix Abscess; Acute Appendicitis With Rupture
Keywords: Acute Appendicitis; Complicated Acute Appendicitis; Uncomplicated Acute Appendicitis; HALP Score
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complicated acute appendicitis cases: Acute appendicitis cases with pathological diagnosis of gangrenous, phlegmonous, perforated or presence of perforation, abscess or plastron in surgical exploration
  Interventions: Procedure: Appendectomy; Diagnostic Test: blood sampling
- Uncomplicated acute appendicitis cases: Acute appendicitis cases without pathological diagnosis of gangrenous, phlegmonous, perforated or presence of perforation, abscess or plastron in surgical exploration
  Interventions: Procedure: Appendectomy; Diagnostic Test: blood sampling

INTERVENTIONS:
Procedure: Appendectomy — Appendectomy (Laparoscopic or conventional open surgery)
  Other Names: Laparoscopic Appendectomy; Conventional Open Appendectomy
Diagnostic Test: blood sampling — Blood samples, in the preoperative period, routinely collected from the patients of acute appendicitis cases

SUMMARY:
Acute abdomen is a frequently encountered clinical condition that can be fatal if not diagnosed early. Acute appendicitis is one of the causes of acute abdomen and is the most common clinical condition leading to acute abdomen worldwide. Therefore, early diagnosis is crucial. Delays in diagnosis can lead to the complication of appendicitis and an increase in its complications, further worsening the clinical picture and raising morbidity and mortality rates.

In patients diagnosed with acute appendicitis, distinguishing between complicated and uncomplicated appendicitis is vital for treatment planning. The evaluation of patients' laboratory and radiological findings are widely used methods in clinical practice for this differentiation.

Recent studies have shown the HALP score has become a new prognostic biomarker in the literature, used to predict a range of clinical outcomes in various neoplasms. To date, the HALP score has been used to evaluate outcomes and prognosis in gastric, colorectal, bladder, prostate, and other cancers, as well as in many other diseases.

The purpose of this study is to determine the clinical impact of using the preoperatively calculated HALP score, derived from blood parameters, in the diagnosis, detection, and treatment of complicated acute appendicitis cases in the preoperative period without the need for additional diagnostic methods.

DETAILED DESCRIPTION:
*Aim of the Study Acute abdomen is a frequently encountered clinical condition that can be fatal if not diagnosed early. Numerous diseases can cause acute abdomen, making accurate and rapid diagnosis extremely important. Acute appendicitis is one of the causes of acute abdomen and is the most common clinical condition leading to acute abdomen worldwide.

In a study by Addiss et al., the incidence of acute appendicitis was approximately 233 per 100,000 people. Although slightly more common in males, there is a lifetime risk of about 7%.

Therefore, early diagnosis is crucial. Delays in diagnosis can lead to the complication of appendicitis and an increase in its complications, further worsening the clinical picture and raising morbidity and mortality rates.

The reported incidence of complicated appendicitis and its complications in various studies ranges from approximately 20% to 30%. This significant rate increases the risk of morbidity and mortality. Thus, early diagnosis and treatment of appendicitis are of great importance to prevent the development of complications.

In patients diagnosed with acute appendicitis, distinguishing between complicated and uncomplicated appendicitis is vital for treatment planning. The evaluation of patients' laboratory and radiological findings are widely used methods in clinical practice for this differentiation.

Alongside laboratory and radiological findings, commonly used scoring systems are also available. Among these, the Alvarado scoring system, first described in 1986, is the most frequently used and popular system, and it remains the primary system consulted in patients with a preliminary diagnosis of acute appendicitis.

Beyond the Alvarado score, the Appendicitis Inflammatory Response (AIR) score, a more recently developed system, is also gaining widespread use. Furthermore, scoring systems created using artificial intelligence with current technologies have also been described.

In recent years, a new scoring system, the HALP score, was first developed by Chen et al. to predict the prognosis of gastric carcinomas. This score is calculated as [hemoglobin (g/L) × albumin (g/L) × lymphocytes (/L)] / platelets (/L).

Recent studies have shown the HALP score has become a new prognostic biomarker in the literature, used to predict a range of clinical outcomes in various neoplasms. Its use has become widespread because HALP is a scoring system composed of routinely used parameters, such as platelet and lymphocyte counts, albumin (indicating nutritional status), and hemoglobin (indicating anemic status).

To date, the HALP score has been used to evaluate outcomes and prognosis in gastric, colorectal, bladder, prostate, and other cancers, as well as in many other diseases.

The purpose of this study is to determine the clinical impact of using the preoperatively calculated HALP score, derived from blood parameters, in the diagnosis, detection, and treatment of complicated acute appendicitis cases in the preoperative period without the need for additional diagnostic methods.

* Material-Methods This study was planned as a retrospective study. For this purpose, it was planned to include patients who were diagnosed with acute appendicitis and operated on in Elazığ Fethi Sekin City Hospital General Surgery Clinic between 01.01.2020 and 01.01.2025. Complete blood count (CBC) and biochemistry values of the patients studied in the preoperative period were recorded by retrospective file scanning. Patients will be divided into two groups according to the postoperative pathology results and exploration findings by examining the pathology results and surgery notes recorded in the system, as complicated acute appendicitis (pathological diagnosis of gangrenous, phlegmonous, perforated or presence of perforation, abscess or plastron in surgical exploration) and uncomplicated acute appendicitis (pathological diagnosis of acute appendicitis). Preopartive HALP score levels will be compared between groups. Since the study is planned retrospectively, the sample size will not be calculated.
* Data Collection Tools Patients' age, gender, complete blood count (CBC), biochemistry, and pathology data will be evaluated.
* Statistical Analysis Data analysis will be performed using the IBM Statistical Analysis for Social Sciences (SPSS) ver 20 statistical software package. The Shapiro-Wilk test will be conducted to assess the normality of distribution for numerical data. Based on the normality of distribution, either the Student's t-test or the Mann-Whitney U test will be used. Numerical data will be presented as mean ± standard deviation (minimum - maximum values) or median (95% Confidence Interval), depending on their conformity to normal distribution.

For comparing categorical data, the Chi-square analysis or Fisher's exact test will be used. Categorical data will be presented as count (n) and percentage (%). Univariate analysis will be performed to identify factors effective in the preoperative prediction of complicated acute appendicitis, followed by multivariate analysis. A probability value of P<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having undergone surgical treatment for a diagnosis of acute appendicitis (Laparoscopic or conventional open surgery)
* Patients with no missing data in their records

Exclusion Criteria:

* Patients under 18 years of age
* Cases of uncomplicated acute appendicitis diagnosed but treated medically
* Patients with incomplete data
* Those with chronic kidney and liver failure
* Patients with liver diseases such as Wilson's disease or alpha-1 antitrypsin deficiency
* Individuals with hematological malignancies like ALL or AML
* Patients with genetic bleeding disorders such as hemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated diagnosed as acute appendicitis.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Preoperative HALP Score | 2020,01,01-2025,01,01
  Manually calculated HALP score from routinely obtained preoperative blood samples of acute appendicitis cases, can be helpful for preoperatively determining complicated acute appendicitis cases without additional cost.

SECONDARY OUTCOMES:
Preoperative cut off value levels of HALP score to determine complicated acute appendicitis | 2020,01,01-2025,01,01
  Manually calculated preoperative HALP score from CBC results of acute appendicitis cases, it will be determined cut-off values according to ROC analysis for complicated acute appendicitis values.

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirkil C, Karabulut K, Aygen E, Ilhan YS, Yur M, Binnetoglu K, Bulbuller N. Appendicitis scores may be useful in reducing the costs of treatment for right lower quadrant pain. Ulus Travma Acil Cerrahi Derg. 2013 Jan;19(1):13-9. doi: 10.5505/tjtes.2013.88714. PMID 23588973
- [Background] Kirkil C, Yigit MV, Aygen E. Long-term results of nonoperative treatment for uncomplicated acute appendicitis. Turk J Gastroenterol. 2014 Aug;25(4):393-7. doi: 10.5152/tjg.2014.7192. PMID 25254521
- [Background] Bozan MB, Yazar FM, Boran OF, Guler O, Azak Bozan A. Are the immature granulocyte count and percentage important in continue medical treatment in acute appendicitis? A prospective, randomized, and controlled study. Ulus Travma Acil Cerrahi Derg. 2022 Jul;28(7):979-987. doi: 10.14744/tjtes.2021.76307. PMID 35775679
- [Background] Guler O, Bozan MB, Alkan Baylan F, Oter S. The Utility of Immature Granulocyte Count and Percentage on the Prediction of Acute Appendicitis in the Suspected Acute Appendicitis According to the Alvarado Scoring System: A Retrospective Cohort Study. Turk J Gastroenterol. 2022 Oct;33(10):891-898. doi: 10.5152/tjg.2022.21865. PMID 35946881
- [Background] Zhang Y, Zhao YY, Qiao J, Ye RH. Diagnosis of appendicitis during pregnancy and perinatal outcome in the late pregnancy. Chin Med J (Engl). 2009 Mar 5;122(5):521-4. PMID 19323901
- [Background] Addiss DG, Shaffer N, Fowler BS, Tauxe RV. The epidemiology of appendicitis and appendectomy in the United States. Am J Epidemiol. 1990 Nov;132(5):910-25. doi: 10.1093/oxfordjournals.aje.a115734. PMID 2239906
- [Background] Khanapure S, Nagral S, Nanavati AJ. A study of events between the onset of symptoms and hospital admission in patients with acute abdomen. Natl Med J India. 2017 Mar-Apr;30(2):65-68. PMID 28816211
- [Background] Bokemeyer A, Ochs K, Fuhrmann V. [Acute Abdomen: Diagnostic Management]. Dtsch Med Wochenschr. 2020 Oct;145(21):1544-1551. doi: 10.1055/a-1007-4264. Epub 2020 Oct 20. German. PMID 33080641
- [Derived] Ag O, Kutluer N, Ogut MZ, Azak Bozan A, Ebiloglu MF, Gunes B, Ayyildiz H, Bozan MB. The Importance of Preoperatively Calculated Halp Score in Differentiating Complicated Acute Appendicitis in Patients With Acute Appendicitis. World J Surg. 2026 Jan;50(1):121-129. doi: 10.1002/wjs.70160. Epub 2025 Nov 25. PMID 41291390